CLINICAL TRIAL: NCT02358863
Title: A Pilot Study of Molecular Profile-Directed Chemotherapy for Metastatic HER2(-) Esophagogastric Adenocarcinoma
Brief Title: Molecularly Tailored Therapy for Patients With Metastatic Cancer of the Esophagus and Stomach
Acronym: mEGA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues with recruitment.
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0973
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Docetaxel; Capecitabine; Cisplatin; Irinotecan; Platinum; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Standard chemotherapy doublet based on molecular testing using one of the following interventions:
  Modified FOLFOX6 Docetaxel/Capecitabine Cisplatin/Irinotecan Cisplatin/Docetaxel IRI/EPI EPI/Docetaxel Irinotecan/Docetaxel Docetaxel
  Interventions: Drug: Modified FOLFOX6; Drug: Docetaxel/Capecitabine; Drug: Cisplatin/Irinotecan; Drug: Cisplatin/Docetaxel; Drug: IRI/EPI; Drug: EPI/Docetaxel; Drug: Irinotecan/Docetaxel; Drug: Docetaxel

INTERVENTIONS:
Drug: Modified FOLFOX6 — Oxaliplatin 85 mg/m2 IV Day 1 every 14 days Leucovorin 400 mg/m2 IV over 2 hours Day 1 5-FU 400 mg/m2 IV over 2 hours Day 1 5-FU 2400 mg/m2 IV over 46 hours Day 1
  Other Names: Oxaliplatin; Eloxatin; Leucovorin; 5-FU; 5-Flourouracil
Drug: Docetaxel/Capecitabine — Docetaxel 30 mg/m2 IV Days 1 and 8 Capecitabine 825 mg/m2 PO BID Days 1-14
  Other Names: Taxotere; Xeloda
Drug: Cisplatin/Irinotecan — Cisplatin 30 mg/m2 IV Days 1 and 8 every 21 days Irinotecan 65 mg/m2 IV days 1 and 8 every 21 days
  Other Names: Platinum; CPT-11; Camptosar
Drug: Cisplatin/Docetaxel — Cisplatin 75 mg/m2 IV Day 1 every 21 days Docetaxel 75 mg/m2 IV Day 1
  Other Names: Platinum; Taxotere
Drug: IRI/EPI — Irinotecan IV over 90 minutes Days 1 and 8 every 28 days Epirubicin IV over 10-15 minutes Days 1 and 8 every 28 days
  Other Names: Irinotecan; CPT-11; Epirubicin; Camptosar
Drug: EPI/Docetaxel — Docetaxel 75 mg/m2 Day 1 every 21 days Epirubicin 50 mg/m2 IV Day 2
  Other Names: Taxotere; Epirubicin
Drug: Irinotecan/Docetaxel — Irinotecan 120 mg/m2 Day 1 every 21 days Docetaxel 50 mg/m2 IV Day 1
  Other Names: CPT-11; Camptosar; Taxotere
Drug: Docetaxel — Docetaxel 60-100 mg/m2 IV day 1 every 21 days
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to determine whether molecular profile-directed therapy (otherwise known as personalized treatment) can improve the effectiveness of standard chemotherapy combinations for patients with esophagogastric adenocarcinoma. A series of tests will be performed on a sample of tumor; based on the results of these tests, a patient will be assigned to a chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, measurable metastatic esophagogastric adenocarcinoma by RECIST criteria
* Patients who have had surgery or radiotherapy with or without neoadjuvant or adjuvant chemotherapy (the wash-out period will be at least 1 month)
* Patients who are not eligible for resection and are chemotherapy naïve
* Patients with HER2(-) status
* Patients who have tumor deposit(s) that are easily accessible by ultrasound or CT guidance
* Patients must have adequate organ function
* Patients must provide written informed consent

Exclusion Criteria:

* Active concurrent malignancy, other than superficial, non-squamous cell carcinoma of the skin or uterine cervix, within the past three years
* ECOG performance status worse than 2
* Prior oral or intravenous chemotherapy for metastatic disease
* Patients with comorbidities that prevent them from being able to receive the chemotherapy regimen
* cardiac ejection fraction 45% or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Marshall, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Modified FOLFOX6 Docetaxel/Capecitabine Cisplatin/Irinotecan Cisplatin/Docetaxel IRI/EPI EPI/Docetaxel Irinotecan/Docetaxel Docetaxel
  Modified FOLFOX6: Oxaliplatin 85 mg/m2 IV Day 1 every 14 days Leucovorin 400 mg/m2 IV over 2 hours Day 1 5-FU 400 mg/m2 IV over 2 hours Day 1 5-FU 2400 mg/m2 IV over 46 hours Day 1
  Docetaxel/Capecitabine: Docetaxel 30 mg/m2 IV Days 1 and 8 Capecitabine 825 mg/m2 PO BID Days 1-14
  Cisplatin/Irinotecan: Cisplatin 30 mg/m2 IV Days 1 and 8 every 21 days Irinotecan 65 mg/m2 IV days 1 and 8 every 21 days
  Cisplatin/Docetaxel: Cisplatin 75 mg/m2 IV Day 1 every 21 days Docetaxel 75 mg/m2 IV Day 1
  IRI/EPI: Irinotecan IV over 90 minutes Days 1 and 8 every 28 days Epirubicin IV over 10-15 minutes Days 1 and 8 every 28 days
  EPI/Docetaxel: Docetaxel 75 mg/m2 Day 1 every 21 days Epirubicin 50 mg/m2 IV Day 2
  Irinotecan/Docetaxel: Irinote
Period: Overall Study
Arm/Group | Chemotherapy
Started | 13
Completed | 10
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Tumor Size Reduction (Objective Response Rate)
Description: Objective response rate is the sum of partial responses plus complete responses and will be assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 13
Participants | 0

ADVERSE EVENTS:
Arm/Group | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 3/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=13)
Abdominal Pain (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=13)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Alkaline phosphatase increased (Hepatobiliary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Oral Mucositis (General disorders) | 1 (2)
Urinary Urgency (Renal and urinary disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (2)
Hypertension (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes